CLINICAL TRIAL: NCT05116332
Title: Comparing the Variation in Laparoscopic Skills Acquisition in Obstetrics & Gynaecology and General Surgical Trainees. (LAGGS Study)
Brief Title: Comparing the Variation in Laparoscopic Skills Acquisition in Obstetrics & Gynaecology and General Surgical Trainees
Acronym: LAGGS
Status: Completed | Type: Observational
Sponsor: Lancaster University (Other)
Collaborators: East Lancashire Hospitals NHS Trust (Other); British Society for Gynaecological Endoscopy (Unknown); Royal College of Obstetricians and Gynecologists (Other); Association of Surgeons of Great Britain and Ireland (Unknown); KARL STORZ Endoscopy-America, Inc. (Industry); Medtronic (Industry)
Responsible Party: Principal Investigator, Abdulwarith Shugaba, Mr, Lancaster University
Other Study IDs: FHMREC20033
Record Dates: First submitted 2021-09-26; First posted 2021-11-11 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Surgery; Fatigue, Mental; Fatigue; Training Group, Sensitivity; Muscle Strain
MeSH Terms: conditions — Mental Fatigue; Fatigue; Hypersensitivity; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstetrics and Gynaecology (O&G): Trainees from ST3/ST4/ST5 grades (n=11) and ST6/ST7 grades (n=12). As O&G training covers both Obstetrics & Gynaecology curriculums, we will recruit trainees in their final two years of training (i.e. ST6 and ST7) with gynaecology special interest; undertaking at least one gynaecology Advanced Training Skills Modules (ATSM). These include advanced laparoscopic training, open and laparoscopic benign abdomen, urogynaecology, gynaecology-oncology and reproductive medicine.
  To measure musculoskeletal (Electromyography) and cognitive fatigue (Electroencephalography): A total of 10 trainees had these measured; ST3/4/5 (n=5) and ST6/7 (n=5).
- General Surgery (GS): Trainees from ST3/ST4/ST5 (n=11) and senior trainees from ST7/ST8 (n=11).
  To measure musculoskeletal (Electromyography) and cognitive fatigue (Electroencephalography): A total of 10 trainees had these measured; ST3/4/5 (n=6) and ST7/8 (n=4)

SUMMARY:
The investigators postulate that there is a difference in the acquisition of Fundamental Laparoscopic Skills (FLS) between general surgical and Obstetrics & Gynaecology (O&G) trainees. This discrepancy is also likely to influence the musculoskeletal and cognitive fatigue trainees experience within both specialties.

Additionally there is likely to be a discrepancy in the expectations of consultants and trainees on skills perceived to be important at the completion of training (CCT).

This study aims to compare and evaluate the discrepancy in FLS acquisition amongst O&G and GS trainees in order to identify areas for improvements in the training pathway, the associated fatigue experience and highlight the expectations perceived to be required at the completion of training.

DETAILED DESCRIPTION:
Laparoscopic surgery (LS) is widely used for an increasing number of procedures in general surgery and obstetrics and gynecology (O&G). However, the psychomotor skills of laparoscopic surgery can be difficult to develop and trainees pursuing a laparoscopic surgical career often face a steep learning curve. Whilst simulation based training can lead to acquisition of transferrable skills, they are not a substitute for the operating theatre.

In both specialties, obtaining adequate exposure to operative work is a multifaceted challenge for the trainees as well as those involved in designing and delivering surgical training. Amongst other factors, NHS pressures driving service provision, European Working Time Directive (EWTD), loss of firm structures, and the cost of training to the trainees themselves have been identified as factors affecting the quality of surgical training in the UK. This is reflected in annual training surveys highlighting concerns over loss of practical training and experience across both specialties.

Whilst the requirements for CCT for general operative skills in open and laparoscopic surgery are comparable in both specialties, the training pathways defer significantly. GS training is 8 years in duration (CT1, CT2, ST3-ST8), whereas O&G consists of 7 years of specialty training (ST1-ST7). The ST1-ST5 years in O&G is mainly devoted to obstetrics and only those trainees pursuing a gynaecological training pathway undertake an intensive period of surgical training in the last two years of their training. The investigators believe there is also earlier exposure to laparoscopy in GS training with a greater volume of laparoscopic work in comparison to O&G training.

So far there is no direct comparison of O&G and GS training pathways and outcomes in laparoscopic skills.

It is known that greater exposure to laparoscopic training is associated with "muscle memory" and may contribute to reducing the physical and mental stress of the surgeon. The investigators would expect trainees to be more efficient at FLS with more laparoscopic surgery exposure. The measurement of muscular and cognitive fatigue can be regarded as a surrogate marker of exposure to laparoscopy giving further insights into the quality of laparoscopic training between the two training programs.

There is currently no literature to highlight expectations and opinions of consultants or programme directors regarding trainees' skills within GS or O&G in the UK, which the investigators believe to be one of the indicators of training standards.

The objectives of the study include; To compare FLS in O&G and GS trainees at ST3/4/5 and those in their final 2 years [ST7/8(GS) and ST6/7 (O&G)], To compare the musculoskeletal and cognitive fatigue experienced by O&G and GS trainees in performing FLS as a marker of their competence, and to compare the standards of laparoscopic ability expected from trainees by experienced GS and gynecological consultants.

Study design:

This is a prospective comparative study and the investigators will recruit participants from professional membership bodies and the North West health education formerly known as the North West deanery. The study is divided into two parts. In part 1, Consultants and trainees from O&G and GS specialties will be contacted electronically through professional membership bodies (O&G consultants through RCOG/BSGE, GS consultants through ASGBI, O&G trainees through RCOG/BSGE, and GS trainees through ASiT). In addition to the above communication methods, the investigators will consider the use of social media and direct emails to increase the survey response rate. The consultants and trainees will be requested to fill out an online short questionnaire designed to assess trainees perceptions of FLS required at CCT and the consultants' expectations of laparoscopic competencies required by trainees at CCT. These surveys will not include any personal details and will be returned anonymously to the investigators via the survey monkey platform. In the second part, the investigators will recruit trainees from the two specialties via the North West deanery by sending out a centralized email requesting them to volunteer for the FLS tasks. In addition to the above recruitment methods, the investigators will consider the use of social media and direct emails to increase trainee recruitment for the study. Trainees will be able to volunteer their help by replying to a secure email address. Those trainees who respond and meet the inclusion criteria will subsequently be invited to attend a study day to perform four FLS tasks with a choice of 6 days across 3 possible weekends.

On the day, trainees will be asked to fill out another short questionnaire to gather some demographic information and account for potential confounding variables. Personal details from these questionnaires will be separated and a study number will be randomly allocated to both parts of the questionnaires and this number will be written on the trainee's badge which will be used for filling out the task evaluation sheets. A single sheet of paper will allow the investigators recognize the study number against the relevant trainee in case there is a need to contact them at some point. This form will be securely stored in a locked cabinet in an NHS locked office accessible only to the research team.

A sub-selection of trainees will be randomly chosen to have an electromyography (EMG) and electroencephalography (EEG) monitoring whilst performing the tasks.

There are four FLS tasks and they are carried out using validated training models called LASTT (Laparoscopic Skills Training and Testing method) and SUTT-1 (Suturing and knot tying Training and Testing method). LASTT is a wooden model and SUTT-1 is a foam sponge. The tasks are:

1. Laparoscopic Camera Navigation; Laparoscopic camera navigation (LCN) assesses the trainee's ability to navigate a 30 degrees camera using either their dominant hand (DH) or their non-dominant hand (NDH). The task requires the trainee to insert a 10mm 30 degrees optic through the central port of the Szabo box trainer. 14 targets will be dispersed around the LASTT model. Each target contains a large size character (either a large number or a large alphabet letter) and a small size character (either a number or an alphabet letter). The large character can be seen from a panoramic field but the smaller character requires the trainee to zoom in. The trainees will be required to sequentially locate all targets whilst being timed.
2. Hand-eye coordination (HEC); To assess HEC, trainees are assessed on their ability to transfer objects as well as navigate the camera. The trainee is expected to use the dominant hand (DH) to hold grasping forceps and the non-dominant hand (NDH) to hold the camera. The LASTT model will be used to assess this. There will be coloured cylinders of different colours, which the trainees will be required to place in corresponding coloured targets nails.
3. Bimanual co-ordination (BMC); BMC is assessed by measuring the time taken for a trainee to transfer 6 objects between their DH and NDH and position them correctly on the LASTT model. Coloured pins will be transferred from a central location to the corresponding coloured targets. The trainees are expected to identify a coloured pushpin (e.g. red), grasp it by the head with grasping forceps(Johans) using their NDH, then transfer the pin to their DH and grasp the pin by its tail using curved forceps like Maryland. The pushpin then needs to be placed in the corresponding disc of the same colour correctly before moving on to the next coloured pushpin.
4. Suturing and knot placement; All trainees will be shown a video demonstration of laparoscopic suturing and intra-corporeal knotting.

A Suturing and knot tying Training and Testing method (SUTT1) foam pad will be used for assessment of suturing and knot placement. This has 5 rows of dots. For this task, the top 4 rows are used and the 5th row is disregarded. Trainees will be expected to place interrupted sutures between two dots and perform 4 intracorporeal knots with 3 throws. A total of 15 minutes will be allowed for this task and the time taken to complete 4 sutures and 4 knots if performed will be recorded. If the trainee runs out of time, then a total number of sutures +/- knots performed within the 15 minutes will be recorded.

Measurement of EMG and EEG; A random selection of trainees will have wireless electromyography (EMG) and electroencephalography (EEG) monitoring whilst performing the above tasks. As the equipment is wireless, it is anticipated that the trainee's freedom of movement will not be affected by it. EMG activity will be measured in the arm, shoulder, upper and lower back muscles, and the EEG activity of interest will be the alpha wave pattern observed during the activities.

ELIGIBILITY:
Inclusion Criteria:

* General surgery trainees at ST3/ST4/ST5/ST7/ST8 levels
* Obstetrics and Gynaecology (O&G) at ST3/ST4/ST5/ST6/ST7 levels
* Consultants and trainees in general surgery and O&G- For surveys on laparoscopic standards.

Exclusion Criteria:

* Those trainees who have had substantial pre-training experience in laparoscopic surgery such as those who have completed another surgical specialty training, have worked as clinical fellows or specialty doctors with substantial exposure to laparoscopic work will be excluded.
* Those trainees who are currently out of program/training and not doing regular clinical work or those trainees outside the North West deanery will also be excluded.
* For the safety of others, anybody with a positive Covid-19 test, symptoms, or contact with -someone infected with the virus will be excluded.
* Currently out of training (maternity leave, Higher degrees not involving any clinical work)
* Those who have completed another surgical specialty training, have worked as clinical fellows or specialty doctor with significant exposure to operative laparoscopic work.
* Withdrawal of consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 22 trainees from GS and 23 trainees from O&G in the northwest deanery.
  - Obstetrics and Gynaecology (O&G): Junior trainees - ST3/ST4/ST5 (n=11) Senior trainees - ST6/ST7 (n=12)
  - General Surgery (GS): ST3/ST4/ST5 (n=11) ST7/ST8 (n=11)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Average time to complete Fundamental Laparoscopic surgery (FLS) tasks. | Over the duration of the 45 minutes when trainees undertake the FLS tasks
  Mean Time Taken (in minutes: seconds) to perform FLS task

SECONDARY OUTCOMES:
EMG measurements of Maximal Voluntary Contraction (MVC) | Over the duration of the 45 minutes when trainees undertake the FLS tasks
  Observed frequency and amplitude of contractions across muscle groups to establish the musculoskeletal demands (demonstrated as muscle fatigue)
EEG measurements of peak alpha power | Over the duration of the 45 minutes when trainees undertake the FLS tasks
  Alpha spindle duration and amplitude during FLS tasks to measure cognitive fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, Lancashire, United Kingdom

REFERENCES:
- [Derived] Khan ZN, Shrestha D, Shugaba A, Lambert JE, Haslett E, Afors K, Bampouras TM, Subar D, Gaffney C, Clark TJ. What laparoscopic skills are necessary for the certificate of completion of training? A prospective nationwide cross-sectional survey of obstetrics and gynaecology and general surgery trainees and consultants in the UK. BMJ Open. 2025 Mar 29;15(3):e095777. doi: 10.1136/bmjopen-2024-095777. PMID 40157732
- [Derived] Khan ZN, Shrestha D, Shugaba A, Lambert JE, Clark J, Haslett E, Afors K, Bampouras TM, Gaffney CJ, Subar DA. Comparing proficiency of obstetrics and gynaecology trainees with general surgery trainees using simulated laparoscopic tasks in Health Education England, North-West: a prospective observational study. BMJ Open. 2023 Nov 10;13(11):e075113. doi: 10.1136/bmjopen-2023-075113. PMID 37949619